CLINICAL TRIAL: NCT05985174
Title: Role of Neutrophil CD64 and Monocyte HLA-DR Markers in the Dignosis of Neonatal Sepsis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aya Gamal Mostafa, Resident of clinical and chemical pathology department, Sohag university hospital, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-23-07-13MS
Record Dates: First submitted 2023-07-16; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Neonatal Sepsis
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cases (Experimental): Neonates of both sexes included in this study with any suspected case of neonatal sepsis with maternal risk factors , e.g., prolonged labor , premature rupture of membrane (PROM) , maternal intrapartum fever and chorioamnionitis , and neonates with sepsis-related clinical signs :temparature instability , apnea , need for supplemental oxygen , bradycardia , tachycardia , hypotension , hypo
  perfusion , feeding intolerance , and abdominal distension .
  Interventions: Diagnostic Test: CD64 , HLA-DR

INTERVENTIONS:
Diagnostic Test: CD64 , HLA-DR — CD64 is atype of integral membrane glycoprotein , when activated , it increases the neutrophils' potential for phagocytosis and bacterial killing .
  HLA-DR is on the surface of monocyte\macrophages , dendritic cells and plays a crucial role in adaptive immune response

SUMMARY:
Neonatal septicemia remains one of the main causes of neonatal morbidity and mortality . Sepsis which is caused by a dysregulated host response to an infectious trigger leading to a life threatening organ dysfunction was declared by the World Health Organization (WHO) on May 2017 as a global health priority that requires resolution for its prevention , dignosis , and management (Monneret et al., 2019). Despite the advances in perinatal and neonatal sepsis remains high and the outcome is still sever (Chirio et al.,2011) .

HLA-DR is on the surface of monocyte \ macrophages , dendritic cells, and B cells and plays a crucial role in adaptive immune response , More than 30 years ago , researches proved an association between the low level of HLA-DR and the development of sepsis (Cheadle at al .,1991) . A decreased expression of mHLA-DR molecules has been associated with immunoparalysis , which is an inflammatory immune responce that occurs in sepsis .(Pradhan et al.,2016).

ELIGIBILITY:
Inclusion Criteria:

* Neonates of both sexes included in this study with any suspected case of neonatal sepsis with maternal risk factors for sepsis , e.g., prolonged labor , premature rupture of membrane (PROM) , maternal intrapartum fever and chorioamnionitis , and neonates with sepsis-related clinical signs: temperature instability, apnea , need for supplemental oxygen ,bradycardia , tachycardia , hypotension , hypoperfusion , feeding intolerance and abdominal distension ,

Exclusion Criteria:

* are the adminstration of antibiotic therapy prior to admission , birth asphyxia , laboratory finding suggestive of inborn error of metabolism , and congenital anomalies including congenital heart diseases .

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
CD64 from a peripheral blood sample measued by FlowCytometry device . | 12 months
  A cluster of differentiation 64 is a type of intergral membrane glycoprotein , when activated , it increases the neutrophil, potential for phagocytosis and bacterial killing .

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chirico G, Loda C. Laboratory aid to the diagnosis and therapy of infection in the neonate. Pediatr Rep. 2011 Feb 24;3(1):e1. doi: 10.4081/pr.2011.e1. PMID 21647274
- [Background] Ng PC, Lam HS. Diagnostic markers for neonatal sepsis. Curr Opin Pediatr. 2006 Apr;18(2):125-31. doi: 10.1097/01.mop.0000193293.87022.4c. PMID 16601490
- [Background] Vazquez Rodriguez S, Arriaga Pizano LA, Laresgoiti Servitje E, Mancilla Ramirez J, Peralta Mendez OL, Villalobos Alcazar G, Granados Cepeda ML, Hernandez Pelaez MG, Cordero Gonzalez G, Arizmendi Villanueva R, Cruz Ramirez JL, Isibasi A, Lopez Macias C, Flores Romo L, Jimenez Zamudio LA, Cerbulo-Vazquez A. Multiparameter flow cytometry analysis of leukocyte markers for diagnosis in preterm neonatal sepsis. J Matern Fetal Neonatal Med. 2021 Jul;34(14):2323-2333. doi: 10.1080/14767058.2019.1666100. Epub 2019 Sep 19. PMID 31537145
- [Background] Aydin M, Barut S, Akbulut HH, Ucar S, Orman A. Application of Flow Cytometry in the Early Diagnosis of Neonatal Sepsis. Ann Clin Lab Sci. 2017 Mar;47(2):184-190. PMID 28442521